CLINICAL TRIAL: NCT02754479
Title: A Clinical Evaluation of the Treatment of Spider Veins on the Ankles Using a Dual Wavelength Laser Emitting 532 nm and 1064 nm Laser Energy
Brief Title: A Clinical Evaluation of the Treatment of Spider Veins on the Ankles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-16-EV07
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Spider Veins
MeSH Terms: conditions — Telangiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Laser treatments (Experimental): Each subject will receive a combination of 532 nm and/or 1064 nm Nd:YAG laser treatment
  Interventions: Device: Nd:YAG laser

INTERVENTIONS:
Device: Nd:YAG laser — Treatment of lower extremity spider veins
  Other Names: Cutera Excel V

SUMMARY:
To evaluate the safety and effectiveness of the Excel V system for the treatment of lower extremity spider veins on the ankles.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the real-world effectiveness of the 532 nm and 1064 nm Nd:YAG lasers within the Cutera Excel V system for the treatment of lower extremity spider veins, specifically on the ankles, within a clinic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 20 to 75 years of age (inclusive).
2. Fitzpatrick Skin Type I - III.
3. Having spider veins on at least 1 ankle measuring 2.0mm or less in diameter, linear or branching, and red, pink, blue and/or purple in color, as assessed by the investigator.
4. Having spider veins on the ankle that are appropriate for laser treatment, as assessed by the investigator.
5. Subject must be able to read, understand and sign the Informed Consent Form.
6. Subject must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
7. Wiling to have limited sun exposure for the duration of the study, including the follow-up period.
8. Willingness to have digital photographs taken of ankle spider veins and agree to use of photographs for presentation, educational or marketing purposes.
9. Agree not to undergo any other procedure for the treatment of ankle spider veins during the study.

Exclusion Criteria:

1. Fitzpatrick Skin Type IV - VI.
2. Pregnant.
3. Having an infection, dermatitis or a rash in the treatment area.
4. Having significant varicosities or perforator veins.
5. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
6. Systemic use of isotretinoin (Accutane®) within 6 months of study participation.
7. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
8. In the opinion of the investigator, any physical or mental condition which might make it unsafe for the subject to participate in this study or which requires systemic therapy that could interfere with this research study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Stankiewicz, MD FAAD, Principal Investigator — DuPage Medical Group
Locations (1):
- DuPage Medical Group, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser Treatments: Each subject will receive a combination of 532 nm and/or 1064 nm Nd:YAG laser treatment on lower extremity spider veins. Darker colored veins located deeper in the dermis are likely to be treated with the 1064 nm Nd:YAG laser. Lighter colored, smaller veins located more superficially are likely to be treated with the 532 nm laser. The intent of the study was not to compare the level of treatment (e.g 532 nm vs 1064nm)
Period: Overall Study
Arm/Group | Laser Treatments
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Laser Treatments: Each subject will receive a combination of 532 nm \and/or 1064 nm Nd:YAG laser treatment on lower extremity spider veins
Arm/Group | Laser Treatments
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessment of Improvement in Treated Spider Veins on the Ankles
Description: Improvement in treated ankle spider veins at 4 weeks post final laser treatment (compared to baseline) as assessed by a blinded evaluators Physician Global Assessment Scale score (Min=0; 4= Max). Higher Score Indicates Better Outcome.
Time Frame: Four weeks post final laser treatment.
Population: 1 enrolled participant was lost to follow-up prior to receiving treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Laser Treatments: Each subject will receive a combination of 532 nm and/or 1064 nm Nd:YAG laser treatment on lower extremity spider veins.
Arm/Group | Laser Treatments
Number analyzed (Participants) | 3
score on a scale | 3.7 (0.6)

2. Secondary Outcome: Subject Satisfaction With Improvement in Treated Spider Veins on the Ankles
Description: Subject satisfaction with improvement in spider veins on the ankles as assessed using the Subject Satisfaction Assessment scale (Min=1, Max=5) at 4 weeks post final treatment. Higher score indicates better outcome.
Time Frame: Four weeks post final laser treatment
Population: 1 enrolled participant was lost to follow-up prior to receiving treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Laser Treatments
Number analyzed (Participants) | 3
score on a scale | 4.3 (1.2)

ADVERSE EVENTS:
Time Frame: Treatment through 4-weeks post final treatment, up to 6 months
Description: Definition of adverse event and/or serious adverse event, used to collect adverse event information, did not differ from the clinicaltrials.gov.
Arm/Group | Laser Treatments
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Treatments (N=3)
Erythema (Skin and subcutaneous tissue disorders) | 3
Edema (Skin and subcutaneous tissue disorders) | 1
Discomfort (Skin and subcutaneous tissue disorders) | 2
Post Inflammatory Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Darkening of Vessel (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Crusting (Skin and subcutaneous tissue disorders) | 1
Nodule (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No